CLINICAL TRIAL: NCT07070843
Title: Effects of Two Different Eye Care Practices on Eye Complications in Mechanically Ventilated Intensive Care Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Saglik Bilimleri University (Other)
Responsible Party: Principal Investigator, Yildiz Deniz, PhD Student, Istanbul Saglik Bilimleri University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IstanbuSBU
Record Dates: First submitted 2025-06-20; First posted 2025-07-17 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Eye Care; Nursing Care; Intensive Care Unit
Keywords: Critical care nursing; Eye infections; Intensive care units; Nursing care
MeSH Terms: conditions — Eye Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group: Standard Eye Care Group (Experimental): There is no established protocol or guideline for eye care in the intensive care unit where the study will be conducted. Routine eye care involves the use of sterile gauze and sterile saline. During routine suctioning procedures, patients' eyes are not closed. If a patient is unable to achieve full eyelid closure, their eyes are covered with an eye patch or sterile gauze. The Schirmer test will be administered to both eyes on the first day (prior to the first eye care intervention), as well as on the fifth, seventh, and tenth days after eye care is performed. Signs and symptoms of eye infection and chemosis will be evaluated daily after the second eye care procedure. Data for this group will be collected, and the administration and documentation of eye care will be monitored.
  Interventions: Other: Control Group: Standard Eye Care Group
- Intervention Group 1: Eye Care Using an Eye Care Kit (Experimental): Eye care will be performed using an eye care kit. All nursing staff in the intensive care unit will receive training regarding the contents and usage of the kit. Patients in this group will receive eye care solely using the kit, following a 4-times-daily care protocol. For patients with lagophthalmos, eyes will be covered using the eye closure pad provided in the kit. The Schirmer test will be performed on both eyes on the first day prior to the initial eye care intervention, and on the fifth, seventh, and tenth days following eye care, with results recorded. Signs of infection and chemosis will be assessed daily after the second eye care session. Data collection will be done using , and eye care administration will be tracked.
  Interventions: Other: Intervention Group 1: Eye Care Using an Eye Care Kit
- Intervention Group 2: Eye Care According to an Eye Care Protocol (Experimental): All ICU nursing staff will be educated on the eye care protocol. A copy of the protocol will be posted on the doors of the rooms of patients receiving care under the protocol.
  Patients' ocular risk factors will be assessed daily, followed by eye care based on the protocol.
  Changes in ocular condition will be assessed and documented, and ICU physicians will be informed as necessary.
  In cases of incomplete eyelid closure, eyes will be covered upon physician notification.
  Patients will be assessed daily for signs of eye infection and conjunctival edema in accordance with the protocol. If signs of infection or complications occur during the day, they will be marked with a (+) symbol on the form.
  The Schirmer test will be applied on the first day (prior to the initial eye care session) and after eye care on days 5, 7, and 10, with results documented.
  Interventions: Other: Intervention Group 2: Eye Care According to an Eye Care Protocol
- Intervention Group 3: Eye Care Using Both the Eye Care Protocol and the Eye Care Kit (Experimental): ICU nursing staff will be educated on the eye care protocol. A copy of the protocol will be posted on the doors of the rooms of patients receiving this combined care.
  Eye care will be performed using the Eye Care Kit developed by the researchers in accordance with the protocol.
  Patients will be assessed for ocular risk factors daily, and eye care will be provided according to the management guidelines of the protocol.
  In cases of incomplete eyelid closure, the eyes will be covered with physician knowledge.
  Patients will be assessed daily for signs of infection and conjunctival edema as per the protocol. Any signs of infection or complications will be marked with a (+) on the form.
  The Schirmer test will be performed on both eyes before the first eye care session on day 1, and following eye care on days 5, 7, and 10, with results recorded.
  Interventions: Other: Intervention Group 3: Eye Care Using Both the Eye Care Protocol and the Eye Care Kit

INTERVENTIONS:
Other: Control Group: Standard Eye Care Group — There is no established protocol or guideline for eye care in the intensive care unit where the study will be conducted. Routine eye care involves the use of sterile gauze and sterile saline. During routine suctioning procedures, patients' eyes are not closed. If a patient is unable to achieve full eyelid closure, their eyes are covered with an eye patch or sterile gauze. The Schirmer test will be administered to both eyes on the first day (prior to the first eye care intervention), as well as on the fifth, seventh, and tenth days after eye care is performed. Signs and symptoms of eye infection and chemosis will be evaluated daily after the second eye care procedure. Data for this group will be collected, and the administration and documentation of eye care will be monitored.
  Arms: Control Group: Standard Eye Care Group
Other: Intervention Group 1: Eye Care Using an Eye Care Kit — Eye care will be performed using an eye care kit. All nursing staff in the intensive care unit will receive training regarding the contents and usage of the kit. Patients in this group will receive eye care solely using the kit, following a 4-times-daily care protocol. For patients with lagophthalmos, eyes will be covered using the eye closure pad provided in the kit. The Schirmer test will be performed on both eyes on the first day prior to the initial eye care intervention, and on the fifth, seventh, and tenth days following eye care, with results recorded. Signs of infection and chemosis will be assessed daily after the second eye care session. Data collection will be done using , and eye care administration will be tracked.
  Arms: Intervention Group 1: Eye Care Using an Eye Care Kit
Other: Intervention Group 2: Eye Care According to an Eye Care Protocol — * All ICU nursing staff will be educated on the eye care protocol. A copy of the protocol will be posted on the doors of the rooms of patients receiving care under the protocol.
  * Patients' ocular risk factors will be assessed daily, followed by eye care based on the protocol.
  * Changes in ocular condition will be assessed and documented, and ICU physicians will be informed as necessary.
  * In cases of incomplete eyelid closure, eyes will be covered upon physician notification.
  * Patients will be assessed daily for signs of eye infection and conjunctival edema in accordance with the protocol. If signs of infection or complications occur during the day, they will be marked with a (+) symbol on the form.
  * The Schirmer test will be applied on the first day (prior to the initial eye care session) and after eye care on days 5, 7, and 10, with results documented.
  Arms: Intervention Group 2: Eye Care According to an Eye Care Protocol
Other: Intervention Group 3: Eye Care Using Both the Eye Care Protocol and the Eye Care Kit — * ICU nursing staff will be educated on the eye care protocol. A copy of the protocol will be posted on the doors of the rooms of patients receiving this combined care.
  * Eye care will be performed using the Eye Care Kit developed by the researchers in accordance with the protocol.
  * Patients will be assessed for ocular risk factors daily, and eye care will be provided according to the management guidelines of the protocol.
  * In cases of incomplete eyelid closure, the eyes will be covered with physician knowledge.
  * Patients will be assessed daily for signs of infection and conjunctival edema as per the protocol. Any signs of infection or complications will be marked with a (+) on the form.
  * The Schirmer test will be performed on both eyes before the first eye care session on day 1, and following eye care on days 5, 7, and 10, with results recorded.
  Arms: Intervention Group 3: Eye Care Using Both the Eye Care Protocol and the Eye Care Kit

SUMMARY:
This study was designed as a prospective, randomized controlled experimental study aiming to compare different approaches to eye care in intensive care patients receiving mechanical ventilation. In this study, patients receiving mechanical ventilation in the intensive care unit will be randomly assigned to four groups using a simple randomization method:

1. Control Group: Standard Eye Care
2. Intervention Group 1: Eye Care with Eye Care Kit
3. Intervention Group 2: Eye Care According to Eye Care Protocol
4. Intervention Group 3: Eye Care with Both Protocol and Eye Care Kit Research Hypotheses H1: Eye care provided using a care protocol is more effective in preventing the development of complications compared to standard eye care.

H2: Eye care provided using an eye care kit is more effective in preventing the development of ocular complications compared to standard eye care.

H3: The combined use of an eye care kit and a care protocol is more effective in preventing the development of ocular complications compared to using the care protocol alone.

H4: The use of an eye care kit is more effective in preventing the development of ocular complications compared to the use of a care protocol.

DETAILED DESCRIPTION:
Study Design and Methodology

In this study, patients receiving mechanical ventilation support in the intensive care unit will be randomly assigned to four groups using a simple randomization method:

1. Control Group: Standard Eye Care Group There is no established protocol or guideline for eye care in the intensive care unit where the study will be conducted. Routine eye care involves the use of sterile gauze and sterile saline. During routine suctioning procedures, patients' eyes are not closed. If a patient is unable to achieve full eyelid closure, their eyes are covered with an eye patch or sterile gauze.
2. Intervention Group 1: Eye Care Using an Eye Care Kit Eye care will be performed using an eye care kit. All nursing staff in the intensive care unit will receive training regarding the contents and usage of the kit. Patients in this group will receive eye care solely using the kit, following a 4-times-daily care protocol. For patients with lagophthalmos, eyes will be covered using the eye closure pad provided in the kit.
3. Intervention Group 2: Eye Care According to an Eye Care Protocol

   * All ICU nursing staff will be educated on the eye care protocol. A copy of the protocol will be posted on the doors of the rooms of patients receiving care under the protocol.
   * Patients' ocular risk factors will be assessed daily, followed by eye care based on the protocol.
   * Changes in ocular condition will be assessed and documented, and ICU physicians will be informed as necessary.
   * In cases of incomplete eyelid closure, eyes will be covered upon physician notification.
   * Patients will be assessed daily for signs of eye infection and conjunctival edema in accordance with the protocol. If signs of infection or complications occur during the day, they will be marked with a (+) symbol on the form.
4. Intervention Group 3: Eye Care Using Both the Eye Care Protocol and the Eye Care Kit

   * ICU nursing staff will be educated on the eye care protocol. A copy of the protocol will be posted on the doors of the rooms of patients receiving this combined care.
   * Eye care will be performed using the Eye Care Kit developed by the researchers in accordance with the protocol.
   * Patients will be assessed for ocular risk factors daily, and eye care will be provided according to the management guidelines of the protocol, including:
   * In cases of incomplete eyelid closure, the eyes will be covered with physician knowledge.

Patients will be assessed daily for signs of infection and conjunctival edema as per the protocol. Any signs of infection or complications will be marked with a (+) on the form.

Evaluation and Analysis During the study period, all patient groups will be assessed at specific intervals for ocular complications (conjunctival edema, eye infections, and dry eye). The effectiveness of the interventions will be measured accordingly. Clinical observation, the Schirmer test, and necessary laboratory/imaging methods will be used for the assessment of ocular complications.

Inter-group differences will be statistically analyzed based on pre-defined dependent variables. The study aims to evaluate whether the use of the eye care protocol and/or the eye care kit provides superior outcomes compared to standard care in the prevention of complications.

The Schirmer test will be administered to both eyes on the first day (prior to the first eye care intervention), as well as on the fifth, seventh, and tenth days after eye care is performed. Signs and symptoms of eye infection and chemosis will be evaluated daily after the second eye care procedure. Data for all group will be collected, and the administration and documentation of eye care will be monitored.

Study Variables Dependent Variables: Conjunctival edema, eye infections, and dry eye observed in ICU patients.

Independent Variables: Age, gender, diagnosis, comorbidities, Glasgow Coma Scale score, use and type of sedation, use and type of muscle relaxants, use and type of antibiotics, duration of mechanical ventilation, ventilator mode, ambient humidity level, blinking frequency, eyelid closure level, albumin levels, Schirmer test results, and use of the eye care kit.

Sample Size The study population will consist of all patients who are connected to mechanical ventilators for diagnosis, treatment, or follow-up and are admitted to the Anesthesia and Reanimation Intensive Care Units of Kartal Dr. Lutfi Kırdar City Hospital, which operates under the Istanbul Provincial Health Directorate.

To determine the required sample size, a power analysis was conducted using the G*Power software (version 3.1.9.4). The power of the study is expressed as 1-β (where β represents the probability of a Type II error). Based on the Chi-square test for independent groups: Goodness-of-fit tests - Contingency tables, and assuming an effect size of d = 0.58 for the secretion variable, the analysis indicated that a minimum of 39 participants per group is required.

Randomization Method After identifying patients who meet the inclusion criteria, they will be randomly assigned to the intervention and control groups. The randomization process will be conducted using a computer-based random number generator (e.g., Excel's RAND() function or tools such as random.org). This approach ensures independence and balance between groups.

Data Collection Tools Data will be collected using the Patient Identification Form, the Glasgow Coma Scale, the "Eye Care Protocol" developed by Ayfer Hiçerimez in 2024 for intensive care unit (ICU) patients, and the Schirmer Test to assess ocular dryness. Eye care interventions will be implemented based on the "Eye Care Kit Application Procedure" developed by the researcher.

1. Patient Identification Form

   * This form includes descriptive and clinical characteristics of the patient, such as: Age, gender, primary diagnosis, comorbidities, Glasgow Coma Scale (GCS) score, use and type of sedatives and muscle relaxants, use and type of antibiotics, duration and mode of mechanical ventilation, ambient humidity level, blink frequency per minute, degree of lagophthalmos, serum albumin level.
   * It also includes ocular risk factors, such as: Absence or reduction of blink reflex, ocular exposure due to incomplete eyelid closure, requirement for invasive mechanical ventilation, positive end-expiratory pressure (PEEP) level, endotracheal suctioning, tightly secured endotracheal tube, use of sedation, use of specific medications (e.g., antihistamines, corticosteroids, immunosuppressive therapies, atropine), prone positioning and overall patient positioning, presence of respiratory tract infections.
2. Eye Care Protocol The Eye Care Protocol, developed by Ayfer Hiçerimez in 2024 for ICU patients, was designed to evaluate the effectiveness of systematic eye care and includes comprehensive assessment and care of both eyes.

   * The first section of the protocol includes the patient's demographic and clinical characteristics, such as: age, gender, diagnosis, comorbidities, Glasgow Coma Scale (GCS) score, use and type of sedatives and muscle relaxants, use and type of antibiotics, duration and mode of mechanical ventilation, ambient humidity level, blink frequency per minute, degree of lagophthalmos, and serum albumin levels.
   * The second section addresses ocular risk factors, including: absence or reduction of the blink reflex, ocular exposure due to incomplete eyelid closure, need for invasive mechanical ventilation, level of positive end-expiratory pressure (PEEP), endotracheal suctioning, tightly secured endotracheal tube, use of sedation, use of medications (e.g., antihistamines, corticosteroids, immunosuppressive therapies, atropine), prone positioning and general patient positioning, and the presence of respiratory tract infections.
   * The third section focuses on eye care management procedures, including:
   * Hand hygiene
   * Elevating the head of the bed to 30-45 degrees unless contraindicated
   * Implementing infection control precautions
   * Performing eye care four times daily using sterile water
   * Assessing the tightness of the endotracheal tube during each eye care session
   * Ensuring that the eyes of intubated patients are closed during suctioning
   * Using separate sterile materials for each eye to prevent cross-infection
   * Assessing and documenting ocular changes (e.g., redness, secretions, crusting at the eyelid margins, eyelash adhesion, discoloration of the conjunctiva, periorbital and conjunctival edema), and informing the ICU physician as needed
   * The fourth section outlines the signs and symptoms of eye infection, including: redness, discharge, crusting of the eyelid margins, eyelash adhesion, discoloration or opacity of the cornea, and periorbital edema.
   * The fifth section addresses ocular complications, specifically conjunctival edema, that may be observed in ICU patients.
3. Dry Eye Monitoring Form The Schirmer Test is used to evaluate dry eye by utilizing thin filter paper strips measuring 5 mm × 30 mm. Each strip is folded at a 90° angle at one end. The bent end of the test strip is placed into the lower conjunctival sac of the eye, and left in place for 5 minutes. After 5 minutes, the strips are removed and the length of the moistened area is measured in millimeters. If the wetted portion exceeds 10 mm, tear production is considered normal. If the moist area measures less than 5 mm, it is indicative of Dry Eye Syndrome. Measurements must be taken separately for each eye.
4. Eye Care Kit Application Procedure The Eye Care Kit was developed by the researchers and includes: two sterile gauze pads (one for each eye), a single-use 10 ml ampoule of distilled water, a 10 ml syringe, and an eye care pad. Two versions of the kit were prepared: one including a sterile eye occlusion pad, and one excluding it. This distinction was made to prevent unnecessary waste in patients who do not require eye occlusion. The kit content and procedure were developed with input from nine experts, and the form was revised accordingly based on their feedback.
5. Standard Eye Care Record Form This form will be used to document the standard eye care provided in the intensive care unit where the study will be conducted. On each day that care is provided, the responsible nurse will complete the form, and the patient will be monitored for a total of ten days. The form was developed based on feedback from nine experts, and necessary revisions were made accordingly.
6. Eye Care Monitoring Form This form will be used to collect data for both the standard eye care group and the eye care kit group.

   * It includes the patient's demographic and clinical characteristics, such as: Age, gender, diagnosis, comorbidities, Glasgow Coma Scale (GCS) score, use and type of sedatives and muscle relaxants, use and type of antibiotics, duration and mode of mechanical ventilation, ambient humidity level, blink frequency per minute, degree of lagophthalmos, and serum albumin level.
   * It also records ocular risk factors, including: Absence or reduction of the blink reflex, ocular exposure due to incomplete eyelid closure, need for invasive mechanical ventilation, positive end-expiratory pressure (PEEP) value, endotracheal suctioning, tightly secured endotracheal tube, use of sedation, medications (e.g., antihistamines, corticosteroids, immunosuppressive therapies, atropine), prone positioning and overall body position, and presence of respiratory tract infections.
   * The monitoring of signs and symptoms of eye infection including redness, discharge, crusting on the eyelid margins, eyelash adhesion, changes in corneal color or loss of corneal transparency, and periorbital edema,
   * The assessment of conjunctival edema,
   * The follow-up of dry eye.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Receiving mechanical ventilation
* Glasgow Coma Scale (GCS) score < 12
* At least 24 hours have passed since ICU admission
* Baseline Schirmer test result indicating tear production > 5 mm prior to study inclusion

Exclusion Criteria:

* Diagnosed with brain death
* Presence of facial or ocular trauma
* Patients with head trauma
* Patients who have undergone brain surgery
* Patients diagnosed with an eye infection or chemosis

Withdrawal Criteria:

* Patient's death during the study period
* Extubation of the patient before completion of the care period

Min Age: 18 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Conjunctival Edema in Critically Ill Patients | Data collection was conducted for 10 consecutive days, beginning 24 hours after admission to the intensive care unit.
  Conjunctival Edema (Chemosis): Chemosis is the edema of the conjunctiva, which is a thin, transparent membrane covering the inner surface of the eyelids and the white part of the eyes (sclera). It refers to the swelling of this membrane that lines the ocular surface.
Ocular Infections in Critically Ill Patients | Data collection was conducted for 10 consecutive days, beginning 24 hours after admission to the intensive care unit.
  Signs and Symptoms of Ocular Infection: Redness, ocular discharge, crusting along the eyelid margins, adhesion of eyelashes (eyelashes sticking together), corneal discoloration (loss of corneal transparency), periorbital edema.
Dry Eye in Critically Ill Patients | Data collection was conducted for 10 consecutive days, beginning 24 hours after admission to the intensive care unit.
  Dry Eye: Dry eye is a multifactorial disease of the ocular surface, defined by tear film instability and associated with symptoms including ocular discomfort, burning sensation, irritation, dryness, visual blurring, and foreign body sensation."

CONTACTS AND LOCATIONS:
Overall Officials: Yildiz Deniz, Principal Investigator — University of Health Sciences (Sağlık Bilimleri Üniversitesi); Besey Oren, Study Director — University of Health Sciences (Sağlık Bilimleri Üniversitesi)
Locations (1):
- University of Health Sciences (Sağlık Bilimleri Üniversitesi), Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results reported in publications derived from this study will be made available to qualified researchers. Shared data will include de-identified datasets and related data dictionaries.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD and related documents will be available starting 6 months after the primary results are published and will remain accessible for up to 5 years from that date.
Access Criteria: Access will be granted to qualified researchers for academic, non-commercial research purposes. Interested researchers must submit a methodologically sound proposal and obtain approval from the study's data access committee. All data will be shared in a de-identified format via secure transfer. The applicant must agree to a data use agreement ensuring data confidentiality and ethical use.